CLINICAL TRIAL: NCT05875584
Title: Exploratory Study of a Novel Based rbcDNA Liquid Biopsy Technique for Colorectal Cancer Early Detection
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Timing Biotech Co.Ltd. (Unknown)
Responsible Party: Principal Investigator, Jun Li, Chief, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: SAHZhejiangU Timing
Record Dates: First submitted 2023-05-04; First posted 2023-05-25 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer; Adenomatous Polyps; Adenoma; Advanced Adenoma
MeSH Terms: conditions — Colorectal Neoplasms; Adenomatous Polyps; Adenoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- advanced adenomas (AA) group: Prospective enrollment of subjects with advanced adenomas
  Interventions: Diagnostic Test: rbcDNA test
- CRC group: Retrospective enrollment of subjects with confirmed colorectal cancer
  Interventions: Diagnostic Test: rbcDNA test

INTERVENTIONS:
Diagnostic Test: rbcDNA test — fecal immunochemical test
  Other Names: FIT

SUMMARY:
Exploration of a novel rbcDNA liquid biopsy technique for early detection of colorectal cancer is a promising development in the field of disease diagnosis and screening. This technique has the potential to establish an efficient and sensitive system for the early detection of colorectal cancer, which can provide a new perspective for individual health monitoring.

DETAILED DESCRIPTION:
Patients who are at high risk of developing colorectal cancer and willing to undergo colonoscopy examination will be asked to collect a stool sample prior to bowel preparation for commercially available FIT (fecal immunochemical test) assay, as well as a blood sample for rbcDNA testing. The colonoscopy and histopathologic examination will be used as a reference for the results obtained from these tests.

ELIGIBILITY:
Inclusion Criteria:

1. Age:40-74Years
2. Sex:All
3. Willing to provide written consent
4. Plan to undergo colorectaloscopy or surgical treatment and be able to provide a complete medical history and cooperate with blood sampling and follow-up visits，other operation.

For advanced adenomas (AA) group:

1. Adenomatous polyps with ≥25% villous component, high-grade dysplasia (HGD), or a diameter ≥10 mm were considered AA. Sessile serrated lesions with diameters ≥10 mm.
2. treatment-naive
3. No other comorbid tumors

For CRC group:

1. Confirmed CRC patients
2. treatment-naive
3. No other comorbid tumors

Exclusion Criteria:

1. Patients with colorectal cancer who have received prior treatment.
2. FAP (familial adenomatous polyposis), Crohn's disease, ulcerative colitis
3. Participants taking anticoagulants such as aspirin or warfarin, or those with coagulation disorders.
4. Prior history of colonoscopy within the past 5 years and removal of lesions
5. Pregnancy or intestinal infarction people
6. Unable to provide informed consent
7. Participants in other clinical trials or who have participated in other clinical trials within 60 days.
8. Unable to provide stool sample and follow-up visits.
9. Presence of major infectious diseases (e.g. HIV, etc.)

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects advanced adenomas and patients with confirmed CRC
Sampling Method: Non-Probability Sample
Enrollment: 598 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Evaluating the sensitivity, specificity, and accuracy of rbcDNA in colorectal cancer screening | Through study completion，an average of 1 year
  A diagnostic colonoscopy procedure is the reference method. Lesions will be confirmed as malignant by histopathologic examination. The rbcDNA test was deployed to a composite score. The tests were processed independently of colonoscopy procedure.

SECONDARY OUTCOMES:
Sensitivity of the rbcDNA screening test with comparison to FIT, with respect to advanced adenoma (AA) and CRC | Through study completion，an average of 1 year
  A diagnostic colonoscopy procedure is the reference method. Lesions will be confirmed as malignant by histopathologic examination. The rbcDNA and FIT test were performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided